CLINICAL TRIAL: NCT06968338
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Ascending Doses of ARGX-213 in Healthy Adult Participants
Brief Title: A Study to Assess the Safety of ARGX-213 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-213-2401
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARGX-213 (Experimental): Participants receiving the experimental drug
  Interventions: Biological: ARGX-213
- Placebo (Placebo Comparator): Participants receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-213 — Intravenous or subcutaneous administrations of ARGX-213
  Arms: ARGX-213
Other: Placebo — Intravenous or subcutaneous administrations of placebo
  Arms: Placebo

SUMMARY:
This study aims to assess the safety of ARGX-213 in healthy adults. Another aim is to measure the amount of ARGX-213 in the blood over time to learn how it moves through the body and acts in the body. The participants will remain in the study for approximately up to 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the local legal age of consent for clinical studies and is aged 18 to 65 years, inclusive, when signing the ICF
* Is a female of nonchild bearing potential (either postmenopausal or surgically sterilized) or a male
* Has a body weight between 50 and 100 kg and a BMI between 18 and 30.5 kg/m^2, inclusive

Exclusion Criteria:

* Has any current or past clinically meaningful medical or psychiatric condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Has a clinically meaningful abnormality detected on ECG recording regarding either rhythm or conduction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, serious adverse events, and adverse events leading to the discontinuation | Up to 17 weeks

SECONDARY OUTCOMES:
ARGX-213 serum concentrations | Up to 17 weeks
Percent change from baseline in total IgG concentrations in serum | Up to 17 weeks
Incidence of antidrug antibodies against ARGX-213 in serum | Up to 17 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No